CLINICAL TRIAL: NCT01384981
Title: Effects of Non-invasive Ventilation on Exercise Capacity and Quality of Life in COPD-patients GOLD III/IV
Brief Title: Effects of Non-invasive Ventilation on Rehabilitation Outcome in COPD-patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: major problems in recruiting patients due to very strict inclusion criteria
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Dr. med Klaus Kenn, Head physician, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGL NIV
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary rehabilitation; COPD; non invasive ventilation; NIV; exercise capacity; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pulmonary rehabilitation with NIV (Active Comparator): Patients receiving nocturnal non-invasiv Ventilation during a 3-week pulmonary Rehabilitation program.
  Interventions: Procedure: pulmonary rehabilitation
- pulmonary rehabilitation without NIV (Sham Comparator): Patients receiving no nocturnal non-invasiv Ventilation during a 3-week pulmonary Rehabilitation program.
  Interventions: Procedure: pulmonary rehabilitation

INTERVENTIONS:
Procedure: pulmonary rehabilitation

SUMMARY:
The aim of the study is to find out if nocturnal non-invasive ventilation during pulmonary rehabilitation increases exercise capacity and quality of life more than pulmonary rehabilitation alone.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of COPD in stages GOLD III/ IV
* receiving optimized medical treatment and long term oxygen therapy if needed
* patients consent to participate in this trial
* no treatment with NIV in the last 4 weeks
* treatment with NIV in the last 4 weeks due to an acute exacerbation

Exclusion Criteria:

* treatment with NIV in the last 4 weeks (except due to an acute exacerbation)
* Intolerance to perform NIV
* Acute exacerbation at baseline or during PR
* Hypercapnia > pCO2 55mmHg
* Inability to perform a 6 minute walking test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
change in 6 minute walking distance | day 1 and 25
  change in 6 minute walking distance from baseline to day 25

SECONDARY OUTCOMES:
change in quality of life (chronic respiratory questionnaire, CRQ) | day 1 and 25
  change in CRQ-Score from baseline to day 25
change quality of life (Saint George´s Respiratory Questionnaire, SGRQ) | day 1 and 25
  change in SGRQ-Score from baseline to day 25

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany